CLINICAL TRIAL: NCT01417936
Title: An Open-label, Single Arm, Phase II Trial to Investigate the Safety and Efficacy of Sym004 in Patients With Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN) Who Have Failed Anti-EGFR Monoclonal Antibody-based Therapy
Brief Title: Sym004 in SCCHN Patients Failing Anti-EGFR Based Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Symphogen A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sym004-02; 2011-000902-24 (EudraCT Number)
Record Dates: First submitted 2011-07-15; First posted 2011-08-16 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-09

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — futuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sym004 (Experimental)
  Interventions: Drug: Sym004

INTERVENTIONS:
Drug: Sym004 — Sym004 will be administered at the dose of 12 milligram per kilogram (mg/kg) as an intravenous infusion every week up to disease progression or withdrawal from treatment.

SUMMARY:
The trial is designed as a multi-center, open label Phase 2 trial that investigates the efficacy and safety of Sym004 in subjects with squamous cell cancer of the head and neck (SCCHN). Subjects included must have responded to previous anti-epidermal growth factor receptor (anti-EGFR) monoclonal antibody-based therapy and subsequently become resistant to that therapy. It is believed that Sym004 has the potential to induce tumor responses and provide a superior treatment option to subjects with advanced SCCHN.

Symphogen was the sponsor for planning/conducting and reporting results for this trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis initially or at relapse of SCCHN of the oral cavity, oropharynx, hypopharynx or larynx
* Recurrent and/or metastatic SCCHN not amenable to curative treatment with surgery and/or (chemo)radiation
* Previous treatment with an anti-EGFR monoclonal antibody (mAb) in the palliative setting either as monotherapy or in combination with chemotherapy or radiotherapy and showing:

  * Documented clinical benefit or response for at least 8 weeks (PR, CR or SD) on the anti-EGFR mAb-based therapy and
  * Documented disease progression (verified by computed tomography [CT] scan or magnetic resonance imaging [MRI] according to RECIST (1.1) during or within 12 weeks following the last administration of anti-EGFR mAb
* Accessible tumor for biopsy and subject acceptance of repeat tumor biopsies
* Other protocol-defined inclusion criteria could apply

Exclusion Criteria:

* More than 2 lines of prior chemotherapy in the palliative setting
* Expected survival <12 weeks
* Subjects with known brain metastases
* Chemotherapy or radiation therapy within 21 days prior to Visit 2 at the exception of palliative radiotherapy for bleeding or pain, which is allowed anytime, if not given on target lesions
* Anti-EGFR mAbs within 14 days prior to Visit 2
* Major surgery within 4 weeks prior to Visit 2 and subjects must have recovered from effects of major surgery
* Other protocol-defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Horak, MD, FACP, Study Director — Symphogen A/S
Locations (10):
- Belgium (3):
  - 3203; Antwerp University Hospital; Department of Medical Oncology, Antwerp, Edegem
  - 3202; Jules Bordet Institute; Clinique d'Oncologie Médicale, Brussels
  - 3201; Cliniques Universitaires St-Luc; Centre du Cancer, Brussels
- 3303; Centre Alexis Vautrin; Département d'Oncologie Médicale, Nancy, Vandoeuvre Les Nancy, France
- Germany (6):
  - 4905; Charité Campus Benjamin Franklin; Hematology, Oncology and Transfusion Medicine, Berlin
  - 4901; Universitätsklinikum Essen, Essen
  - 4904; Universitätsklinikum Freiburg, Freiburg im Breisgau
  - 4906; University Medical Center Hamburg Eppendorf; Department of Otorhinolaryngology and Head and Neck Surgery, Hamburg
  - 4907; University Hospital Heidelberg; Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
  - 4902; University of Leipzig, Leipzig

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Machiels JP, Specenier P, Krauss J, Dietz A, Kaminsky MC, Lalami Y, Henke M, Keilholz U, Knecht R, Skartved NJ, Horak ID, Pamperin P, Braun S, Gauler TC. A proof of concept trial of the anti-EGFR antibody mixture Sym004 in patients with squamous cell carcinoma of the head and neck. Cancer Chemother Pharmacol. 2015 Jul;76(1):13-20. doi: 10.1007/s00280-015-2761-4. Epub 2015 May 8. PMID 25952795

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject (informed consent): 15 July 2011. Last subject completed: 08 October 2012; Clinical data cut-off: 08 October 2012. Subjects randomized at 10 centers in Belgium, France and Germany.
Pre-assignment Details: A total of 28 subjects were screened for eligibility, 2 were excluded (mainly non-fulfillment of inclusion or exclusion criteria) and 26 subjects were randomized.
Groups:
- Sym004: Sym004 was administered at the dose of 12 milligram per kilogram (mg/kg) as an intravenous infusion every week up to disease progression or withdrawal from treatment.
Period: Overall Study
Arm/Group | Sym004
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) comprised all subjects who had been exposed to trial drug irrespective of their compliance to the planned course of treatment.
Arm/Group | Sym004
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Time
Description: The PFS time was defined as the time from first infusion of Sym004 until progressive disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. or death. PD was defined as at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on trial. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm). The unequivocal progression of existing non-target lesions and the appearance of one or more lesions was also considered progression. Subjects who died without confirmed PD were considered as progressed. Subjects who died or showed PD more than 21 days after last treatment were censored (that is, were considered alive without progression on Day 21 after last treatment). Evaluation was done using Kaplan-Meier estimates.
Time Frame: Time from the first infusion of Sym004 until progressive disease or death, assessed up to 24 weeks
Population: The FAS comprised all subjects who had been exposed to trial drug irrespective of their compliance to the planned course of treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sym004
Number analyzed (Participants) | 26
days | 82 [41 to 140]

2. Secondary Outcome: Objective Tumor Response and Derived Endpoints (Objective Response Rate and Disease Control Rate)
Description: Best objective tumor response was defined as the occurrence of complete response (CR), partial response (PR), stable disease (SD), or PD according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
  Objective response was defined as the occurrence of CR or PR according to RECIST Version 1.1. Disease control was defined as the occurrence of CR, PR or SD according to RECIST Version 1.1.
  CR: Disappearance of all lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 mm; PR: At least a 30% decrease in the sum of diameters of all - lesions, taking as reference the baseline sum diameters; SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on trial.
Time Frame: Time from first infusion of Sym004 until disease progression or death, assessed up to 18 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Sym004
Number analyzed (Participants) | 26
Percentage of subjects
  CR | 0 [0 to 0]
  PR | 0 [0 to 0]
  SD | 50.0 [29.9 to 70.1]
  PD | 23.1 [9.0 to 43.6]

3. Secondary Outcome: Duration of Overall Response
Description: Duration of overall response was defined as the time from the first time point where measurement criteria are met for CR or PR until first date of recurrence or PD was objectively documented according to RECIST Version 1.1. Duration of overall response was censored at date of last imaging data of measured lesions if no confirmation of recurrence or PD was available.
Time Frame: Time from first infusion of Sym004 until disease progression or death, assessed up to 18 months
Population: Duration of overall response could not be calculated as no subject showed CR or PR.
Arm/Group | Sym004
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Progression (TTP)
Description: The TTP was defined as the time from first infusion of Sym004 until disease progression according to RECIST Version 1.1 criteria. Disease progression was defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. The subjects who died without prior assessment of PD were censored for TTP.
Time Frame: Time from first infusion of Sym04 until disease progression, assessed up to 18 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sym004
Number analyzed (Participants) | 26
days | 85 [42 to 147]

5. Secondary Outcome: Overall Survival Time
Description: Overall survival time was defined as the time from first infusion of Sym004 until date of death. Subjects who withdraw the consent or lost to follow-up were censored.
Time Frame: Time from first infusion of Sym004 until death, assessed up to 18 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sym004
Number analyzed (Participants) | 26
days | 156 [86 to 202]

6. Secondary Outcome: Number of Subjects With Detectable Biomarkers at Any Visit
Description: The biomarkers human papilloma virus (HPV), mutated epidermal growth factor receptor (EGFRvIII), c-MET and human epidermal growth factor receptor (HER) 2, HER3 were analyzed only in tumor cells while EGFR, phosphorylated epidermal growth factor receptor (pEGFR), and Ki-67 were analyzed both in tumor and skin biopsy cells.
Time Frame: Weeks 0 and 4; and 4 weeks after last dose
Population: The FAS comprised all subjects who had been exposed to trial drug irrespective of their compliance to the planned course of treatment. "n" signifies subjects evaluable for specified biomarker type.
Measure: Number; unit: Subjects
Arm/Group | Sym004
Number analyzed (Participants) | 26
Subjects
  Tumor biopsy: HPV (n=19) | 1
  Tumor biopsy: EGFRvIII (n=21) | 0
  Tumor biopsy: cMET (n=19) | 6
  Tumor biopsy: HER2 (n=17) | 0
  Tumor biopsy: HER3 (n=17) | 0
  Skin biopsy: EGFR (n=18) | 0
  Tumor biopsy: EGFR (n=11) | 0
  Tumor biopsy: pEGFR (n=26) | 0
  Skin biopsy: pEGFR (n=26) | 0
  Skin biopsy: Increase in Ki67 (n=18) | 9
  Skin biopsy: Decrease in Ki67 (n=18) | 9
  Tumor biopsy: Decrease in Ki67 (n=11) | 4

7. Secondary Outcome: Area Under the Serum Concentration Curve From Time Zero to 168 Hours (AUC [0-168])
Description: The AUC (0-168h) was estimated by determining the total area under the curve of the concentration versus time curve.
Time Frame: Pre-treatment, 1, 2, 4, 8, 24, and 48 hours post-infusion at Week 0 and Week 3
Population: The FAS comprised all subjects who had been exposed to trial drug irrespective of their compliance to the planned course of treatment. 'n' signifies subjects who were evaluable at given time points.
Measure: Mean (Standard Deviation); unit: microgram-hour/milliliter
Arm/Group | Sym004
Number analyzed (Participants) | 26
microgram-hour/milliliter
  Week 0 (n=26) | 17574.9 (5863.6)
  Week 3 (n=23) | 25690.8 (14857.1)

8. Secondary Outcome: Area Under the Serum Concentration Curve From Time Zero to Infinity (AUC [0-inf])
Description: The AUC (0-inf) was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity.
Time Frame: Pre-treatment, 1, 2, 4, 8, 24, and 48 hours post-infusion at Week 0 and Week 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: microgram-hour/milliliter
Arm/Group | Sym004
Number analyzed (Participants) | 26
microgram-hour/milliliter
  Week 0 (n=24) | 24620.8 (7883.7)
  Week 3 (n=15) | 61655.7 (22954.9)

9. Secondary Outcome: Maximum Serum Concentration (Cmax)
Time Frame: Pre-treatment, 1, 2, 4, 8, 24, and 48 hours post-infusion at Week 0 and Week 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: microgram/milliliter
Arm/Group | Sym004
Number analyzed (Participants) | 26
microgram/milliliter
  Week 0 (n=26) | 248.4 (82.7)
  Week 3 (n=23) | 299.8 (139.0)

10. Secondary Outcome: Minimum Serum Concentration (Cmin)
Time Frame: Pre-treatment, 1, 2, 4, 8, 24, and 48 hours post-infusion at Week 0 and Week 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: microgram/milliliter
Arm/Group | Sym004
Number analyzed (Participants) | 26
microgram/milliliter
  Week 0 (n=26) | 48.2 (20.1)
  Week 3 (n=23) | 93.6 (45.3)

11. Secondary Outcome: Clearance (CL)
Description: Clearance of a drug was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes.
Time Frame: Pre-treatment, 1, 2, 4, 8, 24, and 48 hours post-infusion at Week 0 and Week 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliliter/hour/kilogram
Arm/Group | Sym004
Number analyzed (Participants) | 26
milliliter/hour/kilogram
  Week 0 (n=24) | 0.55 (0.22)
  Week 3 (n=15) | 0.22 (0.08)

12. Secondary Outcome: Terminal Half Life (T1/2)
Description: The apparent terminal half-life was defined as the time required for the serum concentration of Sym004 to decrease 50% in the final stage of its elimination.
Time Frame: Pre-treatment, 1, 2, 4, 8, 24, and 48 hours post-infusion at Week 0 and Week 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Sym004
Number analyzed (Participants) | 26
hour
  Week 0 (n=24) | 89.1 (26.5)
  Week 3 (n=15) | 140.7 (37.6)

13. Secondary Outcome: Time to Reach Maximum Serum Concentration (Tmax)
Time Frame: Pre-treatment, 1, 2, 4, 8, 24, and 48 hours post-infusion at Week 0 and Week 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Sym004
Number analyzed (Participants) | 26
hour
  Week 0 (n=26) | 6.0 (5.4)
  Week 3 (n=23) | 4.7 (3.4)

14. Secondary Outcome: Time to Reach Minimum Serum Concentration (Tmin)
Time Frame: Pre-treatment, 1, 2, 4, 8, 24, and 48 hours post-infusion at Week 0 and Week 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Sym004
Number analyzed (Participants) | 26
hour
  Week 0 (n=26) | 163.5 (22.9)
  Week 3 (n=23) | 58.4 (81.8)

15. Secondary Outcome: Volume of Distribution (Vz)
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug needed to be uniformly distributed to produce the desired serum concentration of a drug.
Time Frame: Pre-treatment, 1, 2, 4, 8, 24, and 48 hours post-infusion at Week 0 and Week 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliliter/kilogram
Arm/Group | Sym004
Number analyzed (Participants) | 26
milliliter/kilogram
  Week 0 (n=24) | 67.0 (23.2)
  Week 3 (n=15) | 40.9 (10.3)

16. Secondary Outcome: Number of Subjects With Adverse Events (AEs), Serious AEs, AEs Leading to Death and AEs Leading to Discontinuation
Description: An adverse event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Time Frame: From the first dose of study drug administration up to 4 weeks after the last dose of study drug administration
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Sym004
Number analyzed (Participants) | 26
Subjects
  AEs | 26
  SAEs | 20
  AEs Leading to Death | 5
  AEs Leading to Discontinuation | 6

ADVERSE EVENTS:
Time Frame: From the first dose of study drug administration up to 4 weeks after the last dose of study drug administration
Arm/Group | Sym004
Serious Adverse Events (participants affected / at risk) | 20/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sym004 (N=26)
Anaemia (Blood and lymphatic system disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Jejunal perforation (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Death (General disorders) | 1
General physical health deterioration (General disorders) | 2
Device related infection (Infections and infestations) | 1
Herpes zoster ophthalmic (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Urinary tract infection bacterial (Infections and infestations) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Fistula (Musculoskeletal and connective tissue disorders) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Tumor haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Prosthesis implantation (Surgical and medical procedures) | 1
Surgery (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sym004 (N=26)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 16
Pruritus (Skin and subcutaneous tissue disorders) | 13
Dry skin (Skin and subcutaneous tissue disorders) | 12
Erythema (Skin and subcutaneous tissue disorders) | 11
Rash (Skin and subcutaneous tissue disorders) | 8
Skin fissures (Skin and subcutaneous tissue disorders) | 6
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Eczema (Skin and subcutaneous tissue disorders) | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 10
Oedema peripheral (Gastrointestinal disorders) | 6
Face oedema (General disorders) | 4
Asthenia (General disorders) | 3
General physical health deterioration (General disorders) | 3
Mucosal inflammation (General disorders) | 3
Chills (General disorders) | 2
Influenza like illness (General disorders) | 2
Pain (General disorders) | 2
Catheter site erythema (General disorders) | 1
Chest pain (General disorders) | 1
Device leakage (General disorders) | 1
Device occlusion (General disorders) | 1
Local swelling (General disorders) | 1
Pyrexia (General disorders) | 1
Xerosis (General disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 8
Stomatitis (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Aphthous stomatitis' (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Lip oedema (Gastrointestinal disorders) | 1
Lip ulceration (Gastrointestinal disorders) | 1
Folliculitis (Infections and infestations) | 5
Infection (Infections and infestations) | 3
Paronychia (Infections and infestations) | 3
Impetigo (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 2
Wound infection (Infections and infestations) | 2
Abscess jaw (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Dermatitis infected (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Purulence (Infections and infestations) | 1
Sputum purulent (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 13
Decreased appetite (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Infections and infestations) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 7
Coagulopathy (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Dizziness (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Hypotension (Vascular disorders) | 2
Flushing (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hyperaemia (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Peripheral coldness (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2
Jaw fracture (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Conjunctivitis (Eye disorders) | 3
Dry eye (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Aggression (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Weight decreased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Neutrophil count increased (Investigations) | 1
Staphylococcus test positive (Investigations) | 1
White blood cell count increased (Investigations) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Otorrhoea (Ear and labyrinth disorders) | 1
Hyperglycaemia (Endocrine disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other